CLINICAL TRIAL: NCT06699797
Title: Pivotal Clinical Trial Evaluating the Safety and Efficacy of the Fully Implanted Acclaim Cochlear Implant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Envoy Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A200
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Sensori-Neural Deafness; Sensorineural Hearing Loss; Sensorineural Hearing Loss (Disorder); Sensorineural Hearing Loss, Bilateral; Sensorineural Hearing Loss, Profound; Sensorineural Hearing Loss, Severe
Keywords: cochlear implant; fully implanted hearing device
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Acclaim CI (Experimental): Participants who receive the Acclaim CI, or who have the implant procedure attempted.
  Interventions: Device: Acclaim Cochlear Implant

INTERVENTIONS:
Device: Acclaim Cochlear Implant — Participants with the Acclaim CI device will be tested during follow-up with their hearing results compared to baseline (before the device implant procedure).

SUMMARY:
The goal of this clinical trial is to learn if the Acclaim CI works to treat severe to profound sensorineural hearing loss in adults. It was also learn about the safety of the Acclaim CI implant. The main questions it aims to answer are:

* Does the Acclaim CI device help participants hear words better compared to before the implants?
* What medical problems do participants have after the Acclaim CI device was implanted?

Participants will:

* Have the Acclaim CI implanted; and
* Visit the clinical site for checkups and tests at 1-Month, 3-Months, 6-Months, and at 1-year and 2-years after the device has been turned on.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form.
2. Able to understand and comply with the requirements of the Study, including surgery and post-implant rehabilitation.
3. Ability to read, write, comprehend, and speak fluently in English.
4. Post-lingually deafened.
5. 18 years of age or older at the time of informed consent.
6. Good health and absence of significant comorbidities, in the opinion of the Principal Investigator.
7. At least 30 days of experience with appropriate bilaterally fit hearing aids.
8. Ear to be implanted has severe to profound hearing loss defined as pure tone average at 500, 1000, 2000 and 4000 Hz ≥ 70 dB.
9. Contralateral ear has moderately severe to profound hearing loss defined as pure tone average at 500, 1000, 2000 and 4000 Hz ≥ 60 dB.
10. Limited benefit from amplification defined as CNC monosyllabic word recognition ≤ 40% in the ear to be implanted and ≤ 60% in the contralateral ear, in the aided condition.
11. Normal middle ear function based on otoscopy and tympanometry.
12. An accessible cochlear lumen and intact cochlear nerve, and no known lesions on the auditory nerve or auditory central nervous system, on the ear to be implanted confirmed with MRI or CT scan.

Exclusion Criteria:

1. Documented duration of severe to profound hearing loss for 20 or more years.
2. Previous cochlear implantation in either ear.
3. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
4. Active external or middle ear pathology (i.e., infections, tympanic membrane perforation, or ossicular chain issues) in the ear to be implanted at the time of screening or in the past 6 months, that could impact the proper functioning of the device.
5. Known history of chronic eustachian tube dysfunction.
6. Prior surgery in the middle ear, inner ear, neck, or infraclavicular region which is anticipated to prevent proper placement or function of the Acclaim CI.
7. Hearing loss/disorder of retrocochlear origin.
8. Diagnosis of auditory neuropathy.
9. Currently using other active implants that are expected to interfere with the Acclaim CI position or function.
10. Known hypersensitivity to silicone rubber, polyurethane, stainless steel, titanium, platinum, or gold.
11. Known hypersensitivity or contraindications to procedural or post-procedural medications that cannot be adequately managed medically.
12. Pregnancy at the time of Acclaim CI implantation.
13. Known need for MRI or ionizing radiation treatment during Study participation.
14. Unrealistic expectations on the Participant's part regarding the possible benefits, risks, and limitations inherent to the surgical procedure and use of the Acclaim CI, in the Principal Investigator's opinion.
15. Unwillingness or inability to comply with all investigational requirements.
16. Additional conditions that would prevent completion of all Study requirements, in the opinion of the Principal Investigator.
17. Participation in an investigational drug study or another device study within 3 months of the Screening Visit.
18. Previous history of meningitis.
19. Deafness, in the ear to be implanted, due to:

    1. a damaged or absent tympanic membrane,
    2. a damaged or absent middle ear,
    3. an absent cochlea,
    4. lesions on the acoustic nerve, or
    5. lesions on the central auditory pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
In the Safety Set, frequency and severity of device and procedure related adverse events, including device deficiencies, reported through 12-Month post-activation | From consent to the 1-year follow-up visit
In the Full Analysis Set, within-subject difference between CNC word score obtained at 12-months post-activation in the Acclaim Only condition and the pre-operative aided score in the ear to be implanted | From consent to the 1-year follow-up visit

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Center for Neurosciences Ear and Hearing Center, Tucson, Arizona
  - Shohet Ear Associates, Seal Beach, California
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Hearts for Hearing, Oklahoma City, Oklahoma
  - MUSC Health, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided